CLINICAL TRIAL: NCT04761354
Title: Characteristics Predicting Clinically Relevant Reduction of Hypertension Following Adrenalectomy for Primary Aldosteronism: a Multicenter Analysis
Brief Title: Predicting Reduction of Hypertension After Adrenalectomy for Primary Aldosteronism: a Multicenter Analysis
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: University of California, San Francisco (Other); Northwestern Memorial Hospital (Other); Weill Medical College of Cornell University (Other); Columbia University (Other); University of Chicago (Other); M.D. Anderson Cancer Center (Other); Boston Medical Center (Other); University Health Network, Toronto (Other); Montreal General Hospital (Other); University of Sydney (Other); University Medical Center Groningen (Other); Maastricht University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Catholic University of the Sacred Heart (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof. dr. M.R. Vriens, Professor in Endocrine and Oncological Surgery, UMC Utrecht
Other Study IDs: 16-196/C
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism; Primary Aldosteronism Due to Conn Adenoma
Keywords: Primary Aldosteronism; Hyperaldosteronism; Adrenalectomy; Blood Pressure
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (16):
- University Medical Center Utrecht: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- University Medical Center Groningen: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Vu University Medical Center Amsterdam: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- University Medical Center Maastricht: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Academic Medical Center Amsterdam: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Istituto di Semeiotica Chirurgica Roma: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- University of California San Francisco: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Northwestern Memorial Hospital: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Weill Cornell Medical Center: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Columbia University Medical Center: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- University of Chicago Medical Center: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- M.D. Anderson Cancer Center: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Boston Medical Center: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- University Health Network Toronto: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- Montreal General Hospital - McGill University: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy
- University of Sydney: Patients who underwent adrenalectomy for primary aldosteronism in case of an aldosterone-producing-adenoma
  Interventions: Procedure: Unilateral adrenalectomy

INTERVENTIONS:
Procedure: Unilateral adrenalectomy
  Other Names: Endoscopic posterior adrenalectomy

SUMMARY:
Primary aldosteronism (PA) is the excessive endogenous production of the mineralocorticoid aldosterone. Although various rare forms of PA exist, the vast majority of cases are accounted by either an aldosterone-producing adenoma (APA) or bilateral adrenal hyperplasia. During the last decades the prevalence of PA has risen, predominantly due to better awareness of disease. Several studies estimated a prevalence of PA up to 17% in an unselected population of hypertensive patients. However, in a population with resistant hypertension the reported prevalence is even higher: 17-23%. This emphasizes the clinical impact of PA on morbidity and mortality due to high blood pressure. Since both hypertension and aldosteronism are independent risk factors for cardiovascular morbidity, the aim of treatment is curation or reduction of both.

After an adrenalectomy for APA normalization of biochemical abnormalities is achieved in almost all cases. Nevertheless, curation of hypertension (systolic blood pressure <140 and diastolic blood pressure <90 mmHg) without the need of antihypertensive medication is accomplished in only 35-45% of the cases. In 2008 the Aldosteronoma Resolution Score (ARS) was developed. This score predicts the likelihood of complete resolution of the hypertension in patients with an aldosteronoma and has been validated by other investigator groups.

Reduction of hypertension is also an important clinical outcome and is reported in 90-98% of the patients after surgery. In most studies reduction is defined as a certain decrease in blood pressure or antihypertensive medication. However, there is no consensus on the precise definition of reduction in these patients, which leads to incomparable results.

The aim of the proposed study is to determine the proportion of patients with clinically relevant reduction of hypertension after adrenalectomy in a large cohort. Furthermore, the investigators aim to determine the characteristics predicting this clinically relevant reduction. Additionally, the investigators evaluate the predictive value of the Aldosteronoma Resolution Score for clinically relevant reduction and aim to develop a scoring system to help clinicians predict the likelihood of reduction of hypertension after adrenalectomy so it can be used for patient counseling.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent unilateral adrenalectomy between 2010 and 2016 for APA.
* Patients with biochemical evidence of primary aldosteronism who underwent adrenalectomy on account of an aldosterone-producing adenoma(APA), proven by Computerized Tomography(CT) or Magnetic Resonance Imaging(MRI) or Adrenal Venous Sampling(AVS).

Exclusion Criteria:

* Age <18 years.
* Missing or incomplete data about preoperative blood pressure and number of antihypertensive drugs.
* Missing or incomplete follow-up data about postoperative blood pressure and number of antihypertensive drugs. We aim enter the blood pressure and number of antihypertensive drugs closest to 6 months after adrenalectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary aldosteronism patients who underwent unilateral adrenalectomy between 2010 and 2016 for APA
Sampling Method: Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2016-03-26 (Actual); Primary Completion 2017-03-26 (Actual); Study Completion 2017-03-26 (Actual)

PRIMARY OUTCOMES:
Postoperative blood pressure measurement | 6 months postoperative
  systolic and diastolic blood pressure via office blood pressure measurements
antihypertensive medication use | 6 months postoperative (corresponding to the entered postoperative blood pressure)
  number of antihypertensives in defined daily dose
resolution of hypertension | 6 months postoperative
  resolution of hypertension score via the PASO consensus criteria

SECONDARY OUTCOMES:
Postoperative serum potassium level | 6 months postoperative
  Serum potassium in mmol/l.
Postoperative plasma aldosterone level in lying and standing position | 6 months postoperative
  Plasma aldosterone in nmol/l.
Postoperative plasma renin activity in lying and standing position | 6 months postoperative
  Plasma renin activity in mg/L/u.
Postoperative aldosterone to renin ratio | 6 months postoperative
  Aldosterone to renin ratio using plasma aldosterone level and plasma renin activity
Postoperative plasma creatinine level | 6 months postoperative
  Plasma creatinine in mg/dL
Pathology | 6 months postoperative
  Final result of pathology after adrenalectomy

CONTACTS AND LOCATIONS:
Overall Officials: Menno R Vriens, MD, Principal Investigator — UMC Utrecht; Gerlof D Valk, MD, Study Director — UMC Utrecht
Locations (14):
- United States (7):
  - University of California San Francisco, San Francisco, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas
- University of Sydney, Sydney, New South Wales, Australia
- Canada (2):
  - University Health Network Toronto, Toronto, Ontario
  - Montreal General Hospital - McGill University, Montreal, Quebec
- Istituto di Semeiotica Chirurgica Roma, Rome, Lazio, Italy
- Netherlands (3):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687
- [Background] Zarnegar R, Young WF Jr, Lee J, Sweet MP, Kebebew E, Farley DR, Thompson GB, Grant CS, Clark OH, Duh QY. The aldosteronoma resolution score: predicting complete resolution of hypertension after adrenalectomy for aldosteronoma. Ann Surg. 2008 Mar;247(3):511-8. doi: 10.1097/SLA.0b013e318165c075. PMID 18376197
- [Background] Utsumi T, Kawamura K, Imamoto T, Kamiya N, Komiya A, Suzuki S, Nagano H, Tanaka T, Nihei N, Naya Y, Suzuki H, Tatsuno I, Ichikawa T. High predictive accuracy of Aldosteronoma Resolution Score in Japanese patients with aldosterone-producing adenoma. Surgery. 2012 Mar;151(3):437-43. doi: 10.1016/j.surg.2011.08.001. Epub 2011 Oct 13. PMID 22000827
- [Background] Aronova A, Gordon BL, Finnerty BM, Zarnegar R, Fahey TJ 3rd. Aldosteronoma resolution score predicts long-term resolution of hypertension. Surgery. 2014 Dec;156(6):1387-92; discussion 1392-3. doi: 10.1016/j.surg.2014.08.019. Epub 2014 Nov 11. PMID 25456916
- [Background] Stowasser M, Gordon RD, Gunasekera TG, Cowley DC, Ward G, Archibald C, Smithers BM. High rate of detection of primary aldosteronism, including surgically treatable forms, after 'non-selective' screening of hypertensive patients. J Hypertens. 2003 Nov;21(11):2149-57. doi: 10.1097/00004872-200311000-00025. PMID 14597859
- [Result] Vorselaars WMCM, Nell S, Postma EL, Zarnegar R, Drake FT, Duh QY, Talutis SD, McAneny DB, McManus C, Lee JA, Grant SB, Grogan RH, Romero Arenas MA, Perrier ND, Peipert BJ, Mongelli MN, Castelino T, Mitmaker EJ, Parente DN, Pasternak JD, Engelsman AF, Sywak M, D'Amato G, Raffaelli M, Schuermans V, Bouvy ND, Eker HH, Bonjer HJ, Vaarzon Morel NM, Nieveen van Dijkum EJM, Vrielink OM, Kruijff S, Spiering W, Borel Rinkes IHM, Valk GD, Vriens MR; International CONNsortium study group. Clinical Outcomes After Unilateral Adrenalectomy for Primary Aldosteronism. JAMA Surg. 2019 Apr 1;154(4):e185842. doi: 10.1001/jamasurg.2018.5842. Epub 2019 Apr 17. PMID 30810749
- [Result] Vorselaars WMCM, van Beek DJ, Postma EL, Spiering W, Borel Rinkes IHM, Valk GD, Vriens MR; International CONNsortium study group. Clinical outcomes after surgery for primary aldosteronism: Evaluation of the PASO-investigators' consensus criteria within a worldwide cohort of patients. Surgery. 2019 Jul;166(1):61-68. doi: 10.1016/j.surg.2019.01.031. Epub 2019 May 1. PMID 31053245
- [Result] Vorselaars WMCM, van Beek DJ, Postma EL, Spiering W, Borel Rinkes IHM, Valk GD, Vriens MR; International CONNsortium Study Group. Validation of the Aldosteronoma Resolution Score Within Current Clinical Practice. World J Surg. 2019 Oct;43(10):2459-2468. doi: 10.1007/s00268-019-05074-z. PMID 31270571
- [Result] Vorselaars WMCM, van Beek DJ, Suurd DPD, Postma E, Spiering W, Borel Rinkes IHM, Valk GD, Vriens MR; International CONNsortium*. Adrenalectomy for Primary Aldosteronism: Significant Variability in Work-Up Strategies and Low Guideline Adherence in Worldwide Daily Clinical Practice. World J Surg. 2020 Jun;44(6):1905-1915. doi: 10.1007/s00268-020-05408-2. PMID 32025781

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT04761354/Prot_SAP_000.pdf